CLINICAL TRIAL: NCT03715088
Title: Impacts of Resistance Training on Acute Secretion of Irisin in Obese Older and Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Responsible Party: Principal Investigator, Martin Senechal, Assistant Professor, University of New Brunswick
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNB Fredericton
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-06

CONDITIONS: Obesity
Keywords: Irisin; Obesity; Resistance Training; Older Adults; Younger Adults; Myokines
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Older Adults (BMI ≥30 kg/m2) (Experimental): Individuals aged 65-75 living with obesity will perform the Resistance Training Intervention.
  Interventions: Behavioral: Resistance Training Intervention
- Younger Adults (BMI ≥30 kg/m2) (Experimental): Individuals aged 18-30 living with obesity will perform Resistance Training Intervention.
  Interventions: Behavioral: Resistance Training Intervention

INTERVENTIONS:
Behavioral: Resistance Training Intervention — Participants will perform 10 different resistance exercises consisting of three sets of 8-10 repetitions, at 80% of 1-RM, separated by 60-second rest intervals between sets. This exercise protocol was chosen based on literature that suggests that the protocol and intensity do not enhance mitochondria biogenesis. Also, it was well tolerated by obese and older individuals.

SUMMARY:
It is established that resistance training improves metabolic health; however, the mechanisms of this process are not fully understood. A biologically active substance, irisin, has recently received interest in the scientific community with respect to its effects on energy expenditure and weight loss. The purpose of this study is to compare the different irisin release response during a resistance exercise training session. The study will compare individuals two different age groups (young adults: age 18-30; older adults: age 65-75) living with obesity.

DETAILED DESCRIPTION:
Background: Worldwide, the number of individuals living with obesity has doubled over the past thirty years. The growing prevalence of obesity is concerning as obesity is known to be one of the main risk factors for many chronic conditions, such as Type 2 diabetes and cardiovascular diseases. Therefore, it is important that the impact of different types of exercise are understood to properly prescribe exercise interventions to individuals living with obesity. Recently, there has been increased interest for a biologically active substances that are secreted during muscle contraction, myokines, regarding their effects on metabolism during exercise. Specifically, a novel myokine, named irisin, has caught the attention of numerous researchers. Irisin has been shown to play an important role in increasing energy expenditure, reducing body weight, and improving glucose metabolism by adipocyte metabolism. As of now, the majority of research has focused on irisin release during endurance activity; however, there is limited research on irisin secretion during resistance exercise training.

Statement of Objectives: The purpose of this pilot study is to first determine whether irisin secretion increases during an acute session of resistance exercise training with obese individuals; and second, to determine whether changes in irisin levels during an acute bout of resistance exercise training can be seen in different age groups for obese individuals.

Methodology: Fifteen young and fifteen old participants will be recruited via advertisement in the local newspaper, on radio stations, and on posters. Inclusion criteria include individuals aged between either 18-30 or 65-75 years old, classified as obese according to their BMI (>30 kg/m2), inactive defined as engaging in less than 150 minutes of moderate to vigorous aerobic exercise, not currently engaged in a resistance exercise training program, no previous diagnosis of Type 2 diabetes, and having no injuries or conditions that would prevent them from performing a resistance exercise training session.

Primary Outcome Measure: The primary outcome measure in this study will be the change in irisin levels during resistance exercise training. A validated enzyme immunoassay kit from Phoenix Pharmaceutical Inc. (EK-067-16) will be used to measure irisin. Our group already has experience with this equipment and these procedures, which has been validated.

Resistance Exercise Session: Participants will come for their first visit at which time they they will perform a test to determine their maximal strength [1-repetition maximal (1-RM)] for each exercise included in the program. During their second visit, participants will perform 10 different resistance exercises consisting of three sets of 8-10 repetitions, at 80% of 1-RM. A 60-second rest will occur between sets. This exercise protocol was selected based on literature that suggests that the protocol and the intensity do not enhance mitochondria biogenesis. Also, this protocol was shown to be well tolerated by obese and older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-35 or 60-75 years old
* Physically inactive (engaging in less than 150 minutes of moderate to vigorous aerobic exercise)
* No previous diagnosis of Type 2 diabetes
* Obese (BMI ≥30kg/m2)

Exclusion Criteria:

* BMI less than 30kg/m2
* History of Type 2 diabetes
* Physically active (engaging in atleast 150 minutes of moderate to vigorous aerobic exercise)
* Injury or condition that prevents performance of resistance training exercise.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Irisin | Baseline (0 minute), 15 minutes, 30 minutes, and 45 minutes during exercise and 45 minutes post exercise
  The primary outcome is the change in irisin during an acute bout of resistance exercise training.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Senechal, PhD, Principal Investigator — University of New Brunswick
Locations (1):
- University of New Brunswick - Kinesiology, Fredericton, New Brunswick, Canada

REFERENCES:
- [Derived] Rioux BV, Brunt KR, Eadie AL, Bouchard DR, Fox J, Senechal M. Impact of acute circuit training on irisin in younger and older overweight adults. Appl Physiol Nutr Metab. 2021 Oct;46(10):1248-1256. doi: 10.1139/apnm-2020-1087. Epub 2021 Apr 22. PMID 33887165